CLINICAL TRIAL: NCT06781281
Title: Neoadjuvant NabPE With or Without Serplulimab for Early-stage Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative (HR+/HER2-) Breast cancer-an Observational Real-world Study.
Brief Title: NabPE With or Without Serplulimab for Early-stage HR+/HER2- Breast Cancer.
Status: Recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Professor, Henan Cancer Hospital
Other Study IDs: HELEN-018RWS
Record Dates: First submitted 2024-12-05; First posted 2025-01-17 (Actual); Last update posted 2025-06-23 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer Invasive
Keywords: HR+/HER2-; PD1; Real-world study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- NabPE+Serplulimab group: Epirubicin 75mg/m2 ivgtt on Day 1+Albumin Paclitaxel 260mg/m2 ivgtt on Day 1+Serplulimab 4.5mg/Kg ivgtt on Day 3, every 3 weeks for 6 cycles.
  Interventions: Drug: Serplulimab; Drug: NabPE
- NabPE: Epirubicin 75mg/m2 ivgtt on Day 1+Albumin Paclitaxel 260mg/m2 ivgtt on Day 1, every 3 weeks for 6 cycles.
  Interventions: Drug: NabPE

INTERVENTIONS:
Drug: Serplulimab — Serplulimab
  Groups: NabPE+Serplulimab group
Drug: NabPE — Epirubicin 75mg/m2 ivgtt +Albumin Paclitaxel 260mg/m2

SUMMARY:
The goal of this clinical study is to learn if serplulimab is effective in early HR+/HER2- breast cancer. This trial serves a prospective parallel control cohort for HELEN-018 (NCT). The main questions it aims to answer are:

Does serplulimab combined with neoadjuvant chemotherapy improve the pCR rate of early HR+/HER2- breast cancer? What medical problems do participants have when receiving serplulimab? Researchers will compare the effect of serplulimab combined with chemotherapy to the effect of chemotherapy reported in literature.

Participants will: Receive serplulimab plus chemotherapy every 3 weeks for 6 cycles; All patients will receive surgery, and the primary end point is a pathological complete response at the time of definitive surgery; After definitive surgery, the participants will receive adjuvant serplulimab every 3 weeks for up to 6 months from the begining of the treatment.

DETAILED DESCRIPTION:
In recent years, significant progress has been made in the immunotherapy of breast cancer, and PD1/PDL1 inhibitors have achieved good results in the treatment of triple-negative breast cancer. There have also been many attempts to apply them in HR+/HER2- breast cancer. In the I-SPY2 study, Pembrolizumab combined with chemotherapy increased the pCR rate of HR+/HER2- breast cancer from 13% in the chemotherapy alone group to 30%. In the KEYNOTE756 study, Pembrolizumab in combination with chemotherapy increased the pCR rate by 8.5% (24.3% vs. 15.6%) compared to the chemotherapy-only arm in HR+/HER2- breast cancer. pCR rates in the nivolizumab arm of the CheckMate 7FL study were 24.5% compared with 13.8% in the control arm. While further long-term follow-up data are still needed to confirm patient benefit, it still provides a new treatment option for HR+/HER2- breast cancer patients.

The neoadjuvant treatment options commonly used for HR+/HER2- breast cancer are mainly anthracycline sequential or combined with paclitaxel chemotherapy regimens. Several clinical studies have confirmed that albumin paclitaxel is more effective than solvent-based paclitaxel, and therefore, albumin paclitaxel in combination with epirubicin has also become a commonly used chemotherapy regimen in clinical practice.

The aim of this study was to explore the efficacy and safety of the Serplulimab combined with nab-paclitaxel and epirubicin in the neoadjuvant treatment of HR+/HER2- breast cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age>=18 years old
2. cT2 - cT4d, or cT1c with axillary lymph node metastasis confirmed clinically and pathologically；
3. Pathologically proven HR+/HER2- breast cancer:

   defined as:
   * positive for ER or PR (IHC nuclear staining >1%)
   * Her-2 negative (IHC 0, 1+ without FISH, or IHC 2+ with no amplification by FISH)；
4. Has clinically measurable lesions:Measurable lesions on ultrasound, mammography, or MR (optional) within 1 month before randomization；
5. Organ and bone marrow function tests within 1 month before chemotherapy suggest no contraindications to chemotherapy；
6. Cardiac ultrasound EF value ≧55%；
7. Females of childbearing age, with a negative serum pregnancy test 14 days before randomization;
8. ECOG score≤1 point;
9. Sign informed consent；

Exclusion Criteria:

1. The patient has evidence of metastatic breast cancer；
2. For this disease, chemotherapy, endocrine therapy, targeted therapy, radiation therapy, etc. have been received;
3. The patient has a second primary malignancy other than adequately treated skin cancer;
4. The patient has been treated with anti-programmed cell death protein 1 (anti-PD-1), anti-programmed death ligand 1 (anti-PD-L1) or anti-PD-L2 drugs, or other immunotherapy；
5. The patient has been diagnosed with immunodeficiency disease or autoimmune disease;
6. The patient has severe lung or heart disease;
7. The patient has active hepatitis B and C;
8. The patient has a history of organ transplantation or bone marrow transplantation;
9. pregnant or breastfeeding women;
10. The investigators considered chemotherapy contraindicated due to serious, uncontrolled other medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All female breast cancer patients diagnosed and scheduled to receive neoadjuvant chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 709 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-11-28 (Estimated); Study Completion 2030-11-28 (Estimated)

PRIMARY OUTCOMES:
pathological complete response | 24 weeks
  After neoadjuvant chemotherapy and surgery, the resected specimen (breast + axilla) was free of any invasive cancer (ie, ypT0/is, ypN0)

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | 5-10 years
  EFS was defined as the time from randomization to any of the following events: disease progression during neoadjuvant therapy, local or distant recurrence, second primary malignancy (breast or other cancer), or death from any cause.
DFS | 5-10 years
  Disease-free Survival,From the date of surgery to the first local, regional, contralateral or distant recurrence, and death from any cause
Objective Response Rate (ORR) | 24 WEEKS
  ORR is defined as the number of target lesion responders as assessed by MRI
adverse events | After each cycle of chemotherapy (21 days as 1 cycle)]
  Evaluate the nature, incidence and severity of chemotherapy adverse events according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Henan cancer hospital, Zhengzhou, China